CLINICAL TRIAL: NCT05730270
Title: Effects of Smartphone-Based Stress Reduction Training on Social Relations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20021623
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Emotions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stress reduction program 1 (Experimental): Participants will complete stress reduction lessons for two weeks
  Interventions: Behavioral: Stress reduction program 1
- Stress reduction program 2 (Experimental): Participants will complete stress reduction lessons for two weeks
  Interventions: Behavioral: Stress reduction program 2
- Waitlist (No Intervention): Participants will have an opportunity to complete one of the two programs of stress reduction lessons after data collection is completed

INTERVENTIONS:
Behavioral: Stress reduction program 1 — Participants will receive daily online lessons
  Arms: Stress reduction program 1
Behavioral: Stress reduction program 2 — Participants will receive daily online lessons
  Arms: Stress reduction program 2

SUMMARY:
The purpose of this research study is to find out how two different online stress reduction training programs affect people's daily experiences and social relations. The researchers think that people's thoughts, emotions, and behavior toward others may be influenced by stress reduction programs. This study will allow them to study the effectiveness of stress reduction programs for important real-world psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Virginia Commonwealth University students
* age 18 years or older
* Healthy
* English literate
* non-immigrant
* not practicing stress reduction techniques for more than 60 minutes a week
* ownership of a smartphone

Exclusion Criteria:

* People who are not Virginia Commonwealth University students
* major, uncorrected sensory impairments and cognitive deficits
* psychiatric disorders or history thereof
* new diagnosis of a (non-acute) medical or psychiatric condition within the last 3 months
* current drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Change in state emotion regulation | Baseline to post intervention, approximately 2 weeks
  Participants will complete a state emotion strategies measure which will ask them to check various actions they are taking to change their thoughts and feelings. Change in total number of actions checked will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States